CLINICAL TRIAL: NCT04708301
Title: Characterisation of Heart Involvement in Fabry Disease With T1 Mapping
Acronym: T1
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2014CD002; REC Reference No. (Other: 14/NW/0064)
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Fabry Disease
Keywords: Fabry disease; Cardiomyopathy; Cardiac Magnetic Resonance Imaging; T1 mapping
MeSH Terms: conditions — Fabry Disease; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biobanking of blood samples for use in future ethically approved research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: T1 mapping — T1 mapping is a specialised heart scan that measures the magnetic properties of heart tissue and displays them as an image or map

SUMMARY:
Fabry disease is a rare lysosomal storage disorder characterised by a genetic deficiency in the α-galactosidase enzyme. This deficiency leads to a progressive accumulation of a fatty substance, called glycosphingolipids within a specific part of our cells called the lysosome. This lysosomal accumulation can have devastating effects on patients with Fabry disease, affecting multiple organs. Heart involvement is particularly feared because it is the leading cause of death in Fabry disease.

Cardiovascular magnetic resonance imaging (cardiac MRI) is a relatively new heart imaging technique. A cardiac MRI technique called T1 mapping can measure the magnetic relaxation properties of heart tissue. T1 mapping is important in Fabry disease because glycosphingolipids have distinct magnetic relaxation properties. The abnormal build up of glycosphingolipid within the heart may be detectable using T1 mapping. This accumulation of glycosphingolipid could identify an earlier form of Fabry disease. Moreover, it is postulated that T1 mapping may inform prognosis and response to therapy.

Whilst promising, further investigation and development of this innovative technique in Fabry disease is required. This study aims to find out more about T1 mapping in Fabry disease. Patients referred for clinical cardiac MRI scanning will also undergo T1 mapping. T1 mapping results will be correlated with other markers of disease severity. This will allow heart muscle T1 to be determined in a larger population of Fabry patients than currently exists in the literature and T1 to be characterised across a wider range of Fabry disease severity than currently exists in the literature.

DETAILED DESCRIPTION:
Anderson-Fabry disease (Fabry disease) is a genetic lysosomal storage disorder. Lysosomes are structures found within cells that contain enzymes which break down waste products and foreign material. In Fabry disease there is an inborn deficiency of an enzyme called α-galactosidase A. This leads to progressive accumulation of a fatty substance, called glycosphingolipid, in the lysosomes.

Accumulation of glycosphingolipid in cells can affect the function of many organs, but in particular it affects the heart, the brain and nerves and the kidneys. It manifests as severe and chronic limb pain, progressive kidney dysfunction, transient ischaemic attacks and strokes, coronary artery disease and heart failure. Heart involvement is particularly important because it is responsible for the majority of deaths in patients with Fabry disease.

Fabry disease affects between 1:17,000 to 1:117,000 people, although the prevalence is likely to be underestimated due to difficulties in diagnosis. It is seen across all ethnic and racial groups. It is a chronic disease with significantly reduced survival (median age of death 50). The culprit gene is carried on the X chromosome, therefore males are generally more severely affected than females, with symptoms beginning in childhood or adolescence. Manifestations are more variable in females, from no apparent disease to full expression, but up to 90% have symptoms.

There is no cure for Fabry disease, however enzyme replacement therapy (ERT), which consists of providing affected patients with the deficient enzyme, is available. ERT has been demonstrated to reverse or slow disease progression before irreversible end-organ damage has occurred. However, there are no uniform guidelines as to which patients should receive ERT, when to start it, how to monitor response and when to stop it. As such, patient care is far from optimal, with patients who would benefit from ERT often getting it too late or potentially not getting it at all. Furthermore, ERT is being started in patients in whom the disease is irreversible, or continued in patients in whom it is no longer of benefit. As well as the implications for patient care, this has significant implications for healthcare provision, given that ERT costs in excess of £100,000 per patient per year.

The reason why there are no good guidelines for ERT is that there is no good test to determine organ involvement or organ response to therapy. As explained above, heart involvement is particularly important but the current technique to assess heart involvement (ultrasound scanning of the heart (echocardiography)) is insensitive to accumulation of glycosphingolipid. Echocardiography allows assessment for heart muscle thickening and impairment of gross pumping function, but such changes occur late and are insensitive for assessing response to ERT. Heart muscle biopsy can determine glycosphingolipid accumulation, however this is very invasive, expensive and not an acceptable technique for this purpose.

A non-invasive technique to detect early heart involvement in Fabry disease, that would guide initiation of ERT, monitor response to ERT and determine which patients will not benefit from ERT, is urgently required, both in terms of improving and individualizing patient care and in terms of optimizing healthcare provision.

Cardiovascular magnetic resonance imaging (cardiac MRI) is a relatively new clinical heart imaging technique. It provides detailed and often unique information about heart structure and function. Cardiac MRI images are acquired using magnetic fields. It is free from ionizing radiation; indeed it is considered to be "one of the safest medical procedures currently available" (www.nhs.uk), and thus is an ideal technique for disease surveillance and treatment monitoring.

One of the unique attributes of cardiac MRI is its ability to non-invasively characterise the make-up of heart muscle tissue. Just like all tissues have mass, all tissues have magnetic properties. A cardiac MRI technique called T1 mapping can measure the magnetic relaxation properties of tissues. T1 mapping techniques have been used to assess other organs for many years, but have only relatively recently been applied to the heart.

Fat has different magnetic properties to heart muscle; specifically it has faster magnetic relaxation than heart muscle. This difference can be measured using T1 mapping - fat has a shorter (or lower value) T1 relaxation time than heart muscle.

As described above, in Fabry disease, there is accumulation of glycosphingolipid in the heart. Also as described, glycosphingolipid is a fatty substance. Therefore, accumulation of this fat in the heart could theoretically be detected using the T1 mapping technique.

Two small studies have demonstrated low T1 mapping values in Fabry disease patients in comparison to healthy volunteers and in comparison to patients with other heart conditions that cause heart muscle thickening (Sado et al Circ Cardiovasc Imaging. 2013;6:392-398 and Thompson et al Circ Cardiovasc Imaging. 2013;6:637-645). Interestingly, low T1 mapping values were seen in the absence of any other detectable changes in heart structure and function, suggesting that this technique could allow early detection of heart involvement in Fabry disease. T1 mapping and other allied cardiac MRI techniques (late gadolinium enhancement and extracellular volume quantification) have also been used to demonstrate heart muscle scarring in Fabry disease, which is irreversible and thus unlikely to be amenable to ERT.

Potentially therefore, cardiac MRI T1 mapping could allow early detection of heart involvement in Fabry disease and thus better guide initiation of ERT, allow monitoring of heart response to ERT and, together with the allied cardiac MRI techniques described, determine when advanced disease is present and thus when ERT should be stopped or is not appropriate to initiate.

Whilst promising, further investigation and development of this innovative technique in Fabry disease is required. This study aims to find out more about T1 mapping in Fabry disease. Patients referred for clinical cardiac MRI scanning will also undergo T1 mapping. T1 mapping results will be correlated with other markers of disease severity. This will allow:

1. Heart muscle T1 to be determined in a larger population of Fabry patients than currently exists in the literature
2. T1 to be characterised across a wider range of Fabry disease severity than currently exists in the literature.

ELIGIBILITY:
Inclusion Criteria:

Patients with Fabry disease Patients attending for a clinical cardiac MRI scan

Exclusion Criteria:

Patients who have a contraindication to cardiac MRI scanning (including pacemakers, defibrillators, intra-ocular metal, prohibitive intracranial aneurysm clips, severe claustrophobia, inability to lie flat).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Fabry disease who are undergoing cardiac MRI scanning as part of their usual clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Myocardial T1 relaxation time | through study completion, an average of 3 years
  T1 time derived from myocardial T1 mapping

SECONDARY OUTCOMES:
Left ventricular ejection fraction | through study completion, an average of 3 years
  Derived from left ventricular volumetric cine imaging
Left ventricular mass | through study completion, an average of 3 years
  Derived from left ventricular volumetric cine imaging
Right ventricular ejection fraction | through study completion, an average of 3 years
  Derived from right ventricular volumetric cine imaging
Myocardial T2 relaxation time | through study completion, an average of 3 years
  T2 time derived from myocardial T2 mapping
Adverse events | Retrospective - data collection to be finalised by the end of February 2021
  Exploratory composite end-point of adverse events during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Univiersty Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided